CLINICAL TRIAL: NCT00915460
Title: An Open-Label Safety Extension Study of AVONEX® (Interferon Beta-1a) Treatment in Subjects Who Completed Biogen Studies C95-812, C96-823, or C97-830
Brief Title: Open-Label Safety Extension Study of Avonex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: C-98-838
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Avonex; Interferon beta-1a; patients at high risk to develop multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Patients previously enrolled in BIogen Idec study C95-812.
  Interventions: Drug: Interferon beta-1a (Avonex)
- 2 (Experimental): Patients previously enrolled in Biogen Idec study C96-823.
  Interventions: Drug: Interferon beta-1a (Avonex)
- 3 (Experimental): Patients previously enrolled in Biogen Idec study C97-830.
  Interventions: Drug: Interferon beta-1a (Avonex)

INTERVENTIONS:
Drug: Interferon beta-1a (Avonex) — dosage and frequency as per Biogen Idec protocol
  Other Names: Avonex

SUMMARY:
To collect data on serious adverse events which occur during extended treatment with Avonex in subjects at high risk for developing multiple sclerosis (MS) and in subjects with secondary progressive MS.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed (as defined below) one of the following Biogen AVONEX® clinical studies and meet the other criteria indicated.
* Subjects enrolled from studies C95-812 and C97-830 must have completed their respective study within 12 months prior to enrollment in C98-838. Subjects enrolled from study C96-823 must have completed the study within 24 months prior to enrollment in C98-838.
* have not been diagnosed with any other disease that accounts for their neurologic symptoms.

Exclusion Criteria:

* History of any significant cardiac, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude therapy with interferon beta.
* History of severe allergic or anaphylactic reactions or history of hypersensitivity to human albumin.
* History of seizure within the 3 months prior to enrollment.
* Abnormal laboratory results at the screening visit:
* History of suicidal ideation or an episode of severe depression within the 3 months prior to enrollment into this study.

Other inclusion and exclusion criteria apply as per Biogen Idec Protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 1999-09; Primary Completion 2003-06 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to collect data on serious adverse events which occur during extended treatment with AVONEX in subjects at high risk for developing MS and in subjects with secondary progressive MS. | The study duration is 7 months

SECONDARY OUTCOMES:
To monitor the occurrence of diagnosed clinically definite multiple sclerosis (CDMS) in subjects who enter this study at high risk for developing MS following an initial demyelinating event. | The study duration is 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Study Director — Biogen